CLINICAL TRIAL: NCT05764148
Title: Effectiveness of Non Face-to-face Behavioral Activation Treatment for Negative Symptoms of Schizophrenia
Brief Title: Effectiveness of Behavioral Activation Treatment for Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inha University Hospital (Other)
Responsible Party: Principal Investigator, Wonhyoung Kim, Associated professor, Inha University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-01-026
Record Dates: First submitted 2023-03-01; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Schizophrenia, Latent; Negative Symptoms in Schizophrenia; Behavioral Activation; Remote Medical Service
Keywords: Schizophrenia; Negative Symptoms in Schizophrenia; behavioral activation; Remote Medical Service
MeSH Terms: conditions — Schizotypal Personality Disorder; Schizophrenia

STUDY DESIGN:
Intervention Model Description: schizophrenia group and treatment as usual
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral activation (Experimental): Behavioral activation
  Interventions: Behavioral: behavioral activation
- Traatment as usual (Placebo Comparator)
  Interventions: Behavioral: behavioral activation

INTERVENTIONS:
Behavioral: behavioral activation — Behavioral Activation (BA) is a specific CBT skill. It can be a treatment all by itself, or can be used alongside other CBT skills such as cognitive restructuring.
  Behavioral activation helps us understand how behaviors influence emotions, just like cognitive work helps us understand the connection between thoughts and emotions.

SUMMARY:
The purpose of this study is to implement a behavior activation remote program for negative symptoms of schizophrenia and to verify whether the behavior activation remote program for negative symptoms of schizophrenia has effects on negative symptoms, cognitive function, and social function of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received a primary diagnosis of schizophrenia
* Patients who are at least 18 years old and under 65 years old
* Patients who show a score of 3 or higher on at least two negative symptom items in the Positive and Negative Syndrome Scale (PANSS)
* The subject selection period is until December 31, 2021, from the IRB approval date.

Exclusion Criteria:

* Patients with a history of organic brain syndrome, epilepsy, or traumatic brain injury
* Patients with comorbidities such as intellectual disability, current alcohol or other substance dependence
* Patients who show a score of 5 or higher on at least two positive symptom items in the Positive and Negative Syndrome Scale (PANSS)
* Patients who have received a diagnosis of major depressive disorder according to the DSM-V criteria by a specialist in psychiatry
* Patients who have received psychological services including components of behavioral activation therapy
* Patients who are at risk of self-harm or harm to others.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
negative function | three month
  improved negative function

SECONDARY OUTCOMES:
cognitive function | three month
  improved cognitive function
depressed mood | three month
  improved depressed mood

CONTACTS AND LOCATIONS:
Locations (1):
- Inha university hospital, Incheon, Jung-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No